CLINICAL TRIAL: NCT04705896
Title: Albumin To Enhance Recovery After Acute Kidney Injury: A Multi-Centre, Randomized, Controlled Trial
Brief Title: Albumin To Enhance Recovery After Acute Kidney Injury
Acronym: ALTER-AKI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); The Kidney Foundation of Canada (Other); The Ottawa Hospital Academic Medical Organization (TOHAMO) Innovation Fund Grant. (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Blood Services (Other); Héma-Québec (Other)
Responsible Party: Principal Investigator, Edward Clark, Principal Investigator, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRF1819
Record Dates: First submitted 2021-01-07; First posted 2021-01-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury; Renal Replacement Therapy; Hypotension; Critical Illness
Keywords: Albumin; Normal Saline; Dialysis; Intensive Care Unit
MeSH Terms: conditions — Acute Kidney Injury; Hypotension; Critical Illness | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with two parallel arms 1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blood Banks at participating sites prepare intravenous hyperoncotic albumin and normal saline (control) in identical infusion mini-bags. Opaque bags and intravenous tubing covers will be used to maintain blinding as much as possible.
  The packaging for normal saline and 25% albumin will be identical (mini-bags) and be covered. The intravenous tubing will have an opaque sleeve to mask any colour discrepancy in the 2 product
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20-25% Albumin fluid (Active Comparator): 100 mL 20-25% Albumin fluid at the initiation of continuous renal replacement therapy (CRRT), prolonged intermittent renal replacement therapy (PIRRT), or intermittent hemodialysis (IHD) and another 100 mL 20-25% Albumin fluid and halfway through RRT sessions in ICU.
  Interventions: Biological: 20-25% Albumin fluid (100 mL)
- Normal Saline (Placebo Comparator): 100 mL at the initiation of CRRT, SLED or IHD and another 100 mL 0.9% Normal Saline halfway through RRT sessions in ICU.
  Interventions: Other: 0.9% Normal Saline (100 mL)

INTERVENTIONS:
Biological: 20-25% Albumin fluid (100 mL) — Participants will be randomized to receive albumin (20-25%) during their RRT sessions (either CRRT, SLED or IHD) in ICU. Once randomized the same fluid will be given for all subsequent RRT sessions for up to 14 days in ICU.
  RRT sessions will be determined as per the treating physician. Boluses will be given at the start of, and halfway through, RRT sessions (i.e. for SLED sessions, at 0 and 4 hours; for IHD sessions, at 0 and 2 hours).
  Arms: 20-25% Albumin fluid
Other: 0.9% Normal Saline (100 mL) — Participants will be randomized to receive normal saline 100 mL boluses during their RRT sessions (either CRRT, SLED or IHD) in ICU. Once randomized the same fluid will be given for all subsequent RRT sessions for up to 14 days in ICU.
  RRT sessions will be determined as per the treating physician. Boluses will be given at the start of, and halfway through, RRT sessions (e.g. for 8 hour SLED sessions, at 0 and 4 hours; for 4 hour IHD sessions, at 0 and 2 hours; for CRRT, after starting/randomization then every 12 hours while continuing on CRRT).
  Arms: Normal Saline

SUMMARY:
Study objectives:

To determine whether, in critically ill patients with Acute Kidney Injury requiring renal replacement therapy (AKI-RRT), randomization to receive intravenous hyperoncotic albumin 20-25% (100 mL X two doses) compared to control/placebo normal saline boluses (100 mL X two doses) given during RRT sessions, leads to:

1. An increase in organ support-free days (primary outcome) at 28 days following randomization; and
2. An increase in RRT-free days (principal secondary outcome) at 28 days following randomization.

DETAILED DESCRIPTION:
Background: Severe Acute Kidney Injury that necessitates renal replacement therapy (AKI-RRT) is a frequent complication of critical illness and portends severe outcomes: high morbidity, an approximately 50% risk of in-hospital death, and increased healthcare resource utilization. Although life-saving when needed, RRT itself may contribute to the poor outcomes associated with AKI-RRT. Since RRT treatments frequently cause hypotension, repeated episodes of kidney and other organ ischemia may occur during RRT. Hypotension during RRT is often triggered by fluid removal. At the same time, there is some evidence that more aggressive ultrafiltration could be beneficial in AKI-RRT.

Albumin is a protein that is the primary contributor to the colloid oncotic pressure maintaining the effective circulating volume (ECV) during RRT. Critically ill patients with AKI-RRT are nearly always hypoalbuminemic. Despite its high cost and limited evidence to support the practice, intravenous hyperoncotic albumin is commonly administered to patients with AKI-RRT in an effort to boost the colloid oncotic pressure and maintain the blood pressure while simultaneously facilitating fluid removal

Objective:

This proposed trial is intended to provide definitive evidence as to the efficacy of a frequently used and expensive intervention to promote hemodynamic stability and augment ultrafiltration during RRT in critically ill patients

Design: A randomized controlled trial with two parallel arms. Setting: The mixed medical-surgical intensive care units of five Canadian tertiary care hospitals with plans to expand to include other centres across Canada and internationally.

Study Population: 856 patients admitted to the Intensive Care Unit (ICU) with AKI requiring treatment with RRT .

Intervention: Participants will be randomized 1:1 to receive either albumin (20-25%) boluses or normal saline placebo boluses at the start and halfway through RRT sessions in ICU, during their RRT treatments to a maximum of 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Admission to a critical care unit/intensive care unit (ICU) for > 24 hours;
* Receiving vasoactive therapy AND/OR undergoing mechanical ventilation (including non-invasive mechanical ventilation (NIMV));
* Immediate initiation of RRT for management of AKI is planned OR additional RRT sessions are imminently planned for patients who already received RRT during their ICU admission;

Exclusion Criteria:

* Initiation of RRT for reasons other than AKI (e.g. drug intoxication, hypothermia) ;
* Known pre-hospitalization end-stage kidney disease;
* Kidney transplant within the past 365 days;
* Presence or clinical suspicion of renal obstruction, rapidly progressive glomerulonephritis, vasculitis, thrombotic microangiopathy or acute interstitial nephritis;
* Advanced cirrhosis (Child Pugh class C [score 10-15]), spontaneous bacterial peritonitis or hepatorenal syndrome;
* Acute peritoneal dialysis used as the initial RRT modality;
* Contraindications to albumin:

  1. Admitted with traumatic brain injury
  2. Increased intra-cranial pressure in those with intra-cranial pressure monitoring
  3. Prior history of anaphylaxis to intravenous albumin
  4. Contraindication or known objection to albumin/blood product transfusions
* Already received 2 or more RRT sessions during ICU admission.
* Limitations of medical therapy precluding RRT/mechanical ventilation/vasoactive medications or plan to transition to palliation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 856 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-08-28 (Estimated); Study Completion 2025-10-23 (Estimated)

PRIMARY OUTCOMES:
Organ-support-free days (OSFD) | 28 days following randomization
  Organ support-free days are defined as days that are both: 1) vasoactive therapy-free; AND 2) mechanical ventilation-free (including NIMV). For patients who die within 28 days following randomization, organ support-free days are counted as -1. An OSFD will be defined as the receipt of < 2 hours of any vasoactive therapy provided by continuous infusion AND the receipt of < 2 hours of either invasive or non-invasive mechanical ventilation, within a 24-hour period.

SECONDARY OUTCOMES:
RRT-free days through day 28 | Through day 28
  For each patient, one point will be given for each calendar day that a patient was free of RRT. For patients who die within 28 days following randomization, RRT-free days are counted as -1.
  An RRT-free day will be defined as a 24-period in which < 2hours of CRRT was received within a 24-hour period and no intermittent RRT sessions were started during the 24-hour period.
Vasoactive therapy free days | Through day 28
  For patients who die within 28 days following initiation of randomization, vasoactive therapy-free days are counted as -1.
  Vasoactive therapy-free days will be defined as receipt of < 2 hours of any vasoactive therapy provided by continuous infusion within a 24-hour period
Mechanical ventilation-free days | Though day 28.
  For patients who die within 28 days following initiation of randomization, mechanical ventilation-free days are counted as -1.
  Mechanical ventilation-free days will be defined as receipt of < 2 hours of either invasive or non-invasive ventilation during a 24-hour period. Invasive mechanical ventilation is that provided via endotracheal tube (including tracheostomy). Noninvasive ventilation will be counted when more than 5 cm H2O of continuous positive airway pressure and more than 5 cm H2O of pressure support when deployed to avoid intubation. Other uses of noninvasive ventilation (eg, chronic nighttime use for chronic obstructive pulmonary disease) will not be counted.
ICU free days | Through 28 days
  For patients who die within 28 days following initiation of randomization, ICU-free days are counted as being -1.
  ICU-free days will be defined as admission to an ICU for < 2 hours within a 24-hour period
Number of participants with death in ICU | Through 28 days
  Mortality within 28 days since randomization
Number of participants with all-cause mortality at 28 days | Through 28 days
  Mortality within 28 days since randomization
Number of participants with all-cause mortality at 90 days | Through 90 days.
  Mortality within 90 days since randomization.
Number of participants with death in ICU, at 28 days, and in-hospital | Through 90 days
  Days from randomization to death in ICU, at 28 days or in-hospital
Number of participants with RRT dependence at 90 days among surviving patients | Through 90 days.
  Defined by the receipt of any form of RRT within +/- 14 days of the 90-day time point following randomization for those alive at 90-days following randomization
Number of participants with composite of death or RRT dependence at 90 days | Through 90 days.
  Defined as death within 90-days following randomization or the receipt of any form of RRT within +/- 14 days of the 90-day time point following randomization
eGFR will be evaluated in all patients alive at Day 90 | At 90 days
  Serum creatinine will be drawn at day 90 (or as close as possible to day 90) and not beyond 132 days after randomization (i.e. we will accept a serum creatinine from Day 90 minus 14 days to Day 90 plus 42 days). eGFR will be derived from the CKD-EPI Creatinine (2021) equation that excludes the race-based coefficient and expressed in mL/min/1.73 m2
Major adverse kidney outcomes, defined as death, RRT dependence, or sustained reduction in kidney function (defined as eGFR < 75% baseline eGFR) at 90 days. | Through 90 days
  eGFR will be derived from the CKD-EPI Creatinine (2021) equation that excludes the race-based coefficient69 and expressed in mL/min/1.73 m2
Hospitalization-free days | Through 90 days.
  Defined as a 24-hour period completely free of an inpatient hospitalization.
EuroQoL EQ-5D-5L which includes a descriptive system (scored from 5 (worst) to 25 (best)) and a visual analogue scale (scored from 0 (worst) to 100 (best)) at day 90. | At 90 days
  Survivors at 90 days will be contacted and evaluated using the EQ-5D-5L which is a measure of health-related quality of life and patient utility
Occurrence of RRT-associated hypotension (for every RRT session in ICU after randomization) | Through 14 days
  Defined as: a drop in blood pressure during RRT requiring initiation or increase in dose of a vasopressor during RRT session or premature discontinuation of RRT session due to hypotension
Daily fluid balance after randomization up until ICU discharge or day 14, whichever comes first | Day 14 or ICU discharge
  Daily net fluid will be calculated based on the medical chart
Difference between ordered and achieved ultrafiltration for all intermittent HD / SLED treatments will be determined according to the medical record up until ICU discharge or day 14, whichever comes first | Day 14 or ICU discharge
  volume will be determined according to the medical record
Daily Sequential Organ Failure Assessment score (SOFA) score after enrollment up until ICU discharge or day 14, whichever comes first | Day 14 or ICU discharge
  The renal component of the SOFA score will be calculated on the basis of urine output only (as all participants will receive RRT and this impacts the creatinine value).
  The GCS score will not be used for the total score (GCS score is difficult is accurately determine in an intubated and sedated participant)
Health Care Costs | Through 365 days.
  An economic evaluation will include the cost of the intervention and control will be assessed using a micro-costing approach,1plus any implications on length of stay, safety events associated with the intervention and/or control, and the costs associated with RRT-dependence up to 365 days following randomizationTo measure these impacts, we will assess hospital and ICU use, physician claims, and subsequent outpatient claims for RRT for all patients within the trial. Consistent with usual practice within a multi-centre clinical trial, valuation of costs will be done for the subset of all patients enrolled within the province of Ontario, Canada (extrapolated based on all patients in the trial) using administrative costing data available from the Institute for Clinical Evaluative Sciences (IC/ES).
Number of alive participants with RRT-dependence at 365 days | Through 365 days
  defined by the patient having a kidney transplant or receipt of any form of RRT within 14 days before or after the 365-days post-randomization time-point
Number of participants with all-cause mortality at 365 days | Through 365 days
  Mortality within 365 days since randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Edward G Clark, MD MSc FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (16):
- Canada (16):
  - The Governors of the University of Calgary, Calgary, Alberta
  - University of Manitoba - Health Sciences Centre, Winnipeg, Manitoba
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Sunnybrook Health Sciences Centre, North York, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Scarborough Health Network, Scarborough Village, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sinai Health System, Toronto, Ontario
  - Lakeridge Health, Whitby, Ontario
  - Centre Integre de Sante et de Services Sociaux de Laval, Laval, Quebec
  - Centre Integre Universitaire de Sante et de Services Sociaux de L'Estrie - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected during the ALTER-AKI trial will be shared with researchers who provide a detailed and methodologically sound proposal, with specific aims. Data sharing will be for the purposes of medical research, with specific data elements provided to answer the research questions in the proposal, and under the auspices of the consent under which the data were originally gathered
Supporting Information: Study Protocol, SAP
Time Frame: Data availability will commence 6 months after the publication of the primary and secondary analyses, with no anticipated end date
Access Criteria: Qualified researchers will need to sign a data sharing and access agreement and will need to confirm that data will only be used for the agreed upon purpose for which data access was granted. The decision to grant access will be made by the trial co-principal investigators, with involvement of the trial steering committee as needed. Proposals to access ALTER-AKI data should be directed to the trial principal investigator via email: Edward Clark--edclark@toh.ca. Costs of preparing and providing partial datasets will be charged to requesting investigators

REFERENCES:
- [Derived] Ullrich EK, Callum J, Clark EG. Use of Intravenous Albumin in Nephrology Practice Should Be Guideline-Based. J Am Soc Nephrol. 2025 Apr 30;36(7):1446-1449. doi: 10.1681/ASN.0000000750. No abstract available. PMID 40305120